CLINICAL TRIAL: NCT03037879
Title: Treating Cognitive Deficits in Traumatic Spinal Cord Injury: A Randomized Clinical Trial
Brief Title: Treating Cognitive Deficits in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEC-16-059
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injury; Blood Pressure; Cerebral Blood Flow; Cognitive Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SPT (Experimental): Speed of Processing Training
  Interventions: Other: SPT
- Control Group SPT (Active Comparator): Control group to SPT treatment group
  Interventions: Other: SPT Control
- mSMT (Experimental): Story Memory Technique
  Interventions: Other: mSMT
- Control mSMT (Active Comparator): Control group to mSMT treatment group
  Interventions: Other: mSMT Control

INTERVENTIONS:
Other: SPT — Participants in the SPT group will receive 10 training sessions over 5 weeks.
  Arms: SPT
Other: SPT Control — Participants in the SPT control group will receive 10 computer-based control sessions over a five-week period during which they will engage in computer-based training. However, they will not be exposed to the training materials central to the SPT.
  Arms: Control Group SPT
Other: mSMT — Participants in the mSMT group will meet with the trainer twice per week for five weeks. Sessions last 45-60 minutes each and are spread over 5 weeks.
  Arms: mSMT
Other: mSMT Control — Participants in the mSMT control group will meet with the therapist at the same frequency and for the same duration as those in the mSMT experimental group. However, subjects will not be exposed to the training materials central to the mSMT.
  Arms: Control mSMT

SUMMARY:
Multiple studies in the spinal cord injury (SCI) population have documented deficits in learning and memory (LM) and processing speed (PS) that adversely impact daily life and the ability to benefit from rehabilitation. The investigators have previously attributed the cognitive deficits demonstrated in the SCI population to low blood pressure (BP) and cerebral blood flow (CBF) and are currently conducting a study to determine the effect of a 30-day elevation in BP (using midodrine hydrochloride - an alpha agonist) on CBF and cognitive performance compared to placebo in hypotensive individuals with SCI. In addition, the investigators believe that cognitive behavior therapy (CBT) may improve cognition independent of changes in BP and CBF in individuals with SCI. The current randomized clinical trial (RCT) will examine the efficacy of 2 treatment protocols shown to be effective in improving cognitive performance in other neurologically impaired populations for use in persons with SCI demonstrating (1) LM impairment and/or (2) PS impairment on objective measures of cognitive functioning during a complete Neuropsychological assessment. Two methods of outcome assessment will be used to examine treatment impact: (1) a traditional Neuropsychological assessment (NP) and (2) an assessment of global functioning (AGF) composed of broader outcome measures that examine the impact of the treatment on everyday life activities. In this way, the investigators will be able to objectively evaluate the presence or absence of changes in memory performance through a NP assessment, while also evaluating the impact of this treatment protocol on everyday life through the AGF. While most studies evaluating the efficacy of cognitive retraining usually employ a pre- and post-training evaluation, such evaluations have been criticized for their lack of ecological validity (i.e., real world generalizability). The present design allows the assessment of the efficacy of these treatment techniques within an SCI population using traditional measures, as well as the assessment of the impact that treatment has on everyday life. The investigators will additionally evaluate the long-term efficacy by including a 6-month post-treatment follow-up. Few studies examine long-term effects, but given the time, labor and expense involved, it is critical to demonstrate long-term efficacy.

DETAILED DESCRIPTION:
104 individuals with SCI will be recruited for eligibility to participate in the study. Participants will be randomly assigned to 4 groups (n=26 per group) story memory technique (mSMT), mSMT control, speed of processing training (SPT) and SPT control.

The study involves 14 visits spread over 8 months. A screening visit, lasting approximately 1 hour. 3 testing sessions lasting 3-4 hours each (Baseline, Immediate and Long-term follow-ups), and 10 intervention sessions that will last approximately 45 minutes each.

Screening: Prior to enrollment in the study protocol, all potential subjects will undergo cognitive screening to determine eligibility for participation.

Baseline: After passing screening, subjects will be scheduled for the baseline evaluation comprised of a cardiovascular/cerebrovascular assessment and cognitive evaluation.

Intervention: Subjects will undergo 10 sessions of training in one of the 4 randomized groups.

Immediate Follow-up Assessment: Subjects will undergo a repeat of the baseline assessments upon completion of the intervention protocol to document changes in PS, LM, BP and CBF following treatment.

Long-Term Follow-up: Subjects will be asked to return to the laboratory 6 months following the intervention for evaluation of the maintenance of the treatment effect over time. Baseline and Immediate follow-up measures of PS, LM, BP and CBF will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Primary language is English;
* Level of Spinal Cord Injury between C1 and T12;
* Non-ambulatory (wheelchair dependent);
* American Spinal Injury Association (AISA) grade A, B or C;
* Spinal Cord Injury occurred more than 1 year ago.

Exclusion Criteria:

* Acute illness or infection.
* Documented history of:
* Controlled or uncontrolled Hypertension or Diabetes Mellitus;
* Stroke;
* Multiple sclerosis & Parkinson's disease;
* Psychiatric disorders (post-traumatic stress disorder, schizophrenia; bipolar disorder);
* Pre-screen MoCA score of < 22 (to rule out dementia);
* Vision impaired - more than 20/60 in worst eye (with prescription eyewear).
* Currently prescribed steroids, benzodiazepines, or neuroleptics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Neuropsychological Tests [Change from baseline at immediate follow up (post treatment) and long term follow-up (6months post treatment)] | Screening (before baseline measures), Baseline, Immediate Follow-up (about 2 months after baseline), Long-term Follow-up (6 months after immediate follow-up)
  NP testing will be conducted to document levels of cognitive performance. NP assessment will identify persons who qualifies for study participation.

SECONDARY OUTCOMES:
Systolic Blood Pressure [Change from baseline at immediate follow up (post treatment) and long term follow-up (6months post treatment)] | Baseline, Immediate Follow-up (about 2 months after baseline), Long-term Follow-up (6 months after immediate follow-up)
  Brachial BP will be measured by a trained technician using a standard adult BP cuff (GE Healthcare Information Technologies, Milwaukee, WI) at 60-second intervals. Beat-to-beat finger arteriolar BP will be monitored continuously from the left middle or ring finger using photoplethysmography (FMS: Finometer, model 2; Amsterdam, Netherlands).
Diastolic Blood Pressure [Change from baseline at immediate follow up (post treatment) and long term follow-up (6months post treatment)] | Baseline, Immediate Follow-up (about 2 months after baseline), Long-term Follow-up (6 months after immediate follow-up)
  Brachial BP will be measured by a trained technician using a standard adult BP cuff (GE Healthcare Information Technologies, Milwaukee, WI) at 60-second intervals. Beat-to-beat finger arteriolar BP will be monitored continuously from the left middle or ring finger using photoplethysmography (FMS: Finometer, model 2; Amsterdam, Netherlands).
Cerebral Blood Flow Velocity [Change from baseline at immediate follow up (post treatment) and long term follow-up (6months post treatment)] | Baseline, Immediate Follow-up (about 2 months after baseline), Long-term Follow-up (6 months after immediate follow-up)
  A transcranial Doppler (TCD) ultrasound probe will be used to locate the left middle cerebral artery (MCA). Once the MCA is located a head harness will be used to secure probe placement for assessment of resting cerebral blood flow velocity (CBFv).

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D., Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided